CLINICAL TRIAL: NCT03581409
Title: Comparison of Dual-Antiplatelet and Triple-Antiplatelet Preparation Using P2Y12 Assay in Patients With High On-Treatment Platelet Reactivity Undergoing Stent-Assisted Coil Embolization for An Unruptured Intracranial Aneurysm
Brief Title: Comparison of Two Different Antiplatelet Preparations for an Unruptured Intracranial Aneurysm
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B-1712/439-001
Record Dates: First submitted 2018-06-14; First posted 2018-07-10 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2019-10

CONDITIONS: Aneurysm, Cerebral; Endovascular Procedures
Keywords: antiplatelet preparation; cerebral aneurysm; coil embolization
MeSH Terms: conditions — Intracranial Aneurysm | interventions — Aspirin; Prasugrel Hydrochloride; Clopidogrel; Cilostazol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- dual-antiplatelet (Experimental): Patients with unruptured aneurysms received dual antiplatelet agents (100 mg of aspirin and 75 mg of clopidogrel) for at least five days before embolization. One day prior to coil embolization, P2Y12 reaction units were measured using VerifyNow. Patients with clopidogrel resistance (greater than 220 PRU) received prasugrel 20mg. After that, dual-antiplatelet (aspirin 100mg & prasugrel 5mg) treatment continued for 3 months through study completion.
  Interventions: Drug: Aspirin; Drug: Prasugrel
- triple-antiplatelet (Experimental): Patients with unruptured aneurysms received dual antiplatelet agents (100 mg of aspirin and 75 mg of clopidogrel) for at least five days before embolization. One day prior to coil embolization, P2Y12 reaction units (PRU) were measured using VerifyNow. Patients with clopidogrel resistance (greater than 220 PRU) received cilostazol 200mg. After that, triple-antiplatelet (aspirin 100mg, clopidogrel 75mg, and cilostazol 200mg) treatment continued for 3 months through study completion.
  Interventions: Drug: Aspirin; Drug: Clopidogrel; Drug: Cilostazol

INTERVENTIONS:
Drug: Aspirin — Aspirin protect tablet
  Other Names: Aspirin protect
Drug: Prasugrel — Prasugrel tablet
  Other Names: Effient
  Arms: dual-antiplatelet
Drug: Clopidogrel — Clopidogrel 75mg tablet
  Other Names: Plavix; Plavitor
  Arms: triple-antiplatelet
Drug: Cilostazol — Cilostazol tablet
  Other Names: Pletaal; Cilostan CR
  Arms: triple-antiplatelet

SUMMARY:
Perform a randomized comparison study of dual-antiplatelet (aspirin, prasugrel) and triple-antiplatelet (aspirin, clopidogrel, and cilostazol) preparation using P2Y12 assay in patients with high on-treatment platelet reactivity undergoing stent-assisted coil embolization for an unruptured intracranial aneurysm

DETAILED DESCRIPTION:
Comparison between dual-antiplatelet and triple-platelet preparation

ELIGIBILITY:
Inclusion Criteria:

* patients with clopidogrel resistance (greater than 220 P2Y12 reaction units using VerifyNow)
* patients with unruptured intracranial aneurysms
* patients over 20 years old
* patients who can communicate with each other
* patients who agreed to this study (with informed consent)

Exclusion Criteria:

* patients with recurrent aneurysms after coiling or clipping
* patients with allergic reaction to antiplatelets
* patients with high risks of hemorrhage
* patients with coagulopathy
* patients with thrombocytopenia (<100,000/mm3)
* patients with liver disease (> 100 of aspartate aminotransferase or alanine aminotransferase)
* patients with renal disease (> 2mg/dL of serum creatinine)
* patients with uncontrolled heart failure or angina
* patients with malignant tumor
* pregnant patients
* patients with past history that may associated with headache, including subarachnoid hemorrhage, head trauma, intracerebral hemorrhage, trigeminal neuralgia, arteriovenous malformation, brain tumor)
* Patients who are determined to be disqualified by researchers

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2021-01-22 (Actual); Study Completion 2021-01-22 (Actual)

PRIMARY OUTCOMES:
Incidence of hemorrhagic complications between 2 arms | through study completion (for 3 months)
  check minor and major hemorrhagic complications of intra- and post-procedures

SECONDARY OUTCOMES:
Change of the level of P2Y12 | through study completion (for 3 months)
  Check the change of the level of P2Y12 according to each arms during study periods
mortality between 2 arms | through study completion (for 3 months)
  check mortality after procedures
Incidence of thromboembolic complications between 2 arms | through study completion (for 3 months)
  check minor and major thromboembolic complications of intra- and post-procedures

CONTACTS AND LOCATIONS:
Overall Officials: Seung Pil Ban, M.D., Study Chair — Seoul National Bundang Hospital
Locations (1):
- Seoul National Univeristy Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Geyik S, Yavuz K, Yurttutan N, Saatci I, Cekirge HS. Stent-assisted coiling in endovascular treatment of 500 consecutive cerebral aneurysms with long-term follow-up. AJNR Am J Neuroradiol. 2013 Nov-Dec;34(11):2157-62. doi: 10.3174/ajnr.A3574. Epub 2013 Jul 25. PMID 23886748
- [Result] Hwang G, Huh W, Lee JS, Villavicencio JB, Villamor RB Jr, Ahn SY, Kim J, Chang JY, Park SJ, Park NM, Jeong EA, Kwon OK. Standard vs Modified Antiplatelet Preparation for Preventing Thromboembolic Events in Patients With High On-Treatment Platelet Reactivity Undergoing Coil Embolization for an Unruptured Intracranial Aneurysm: A Randomized Clinical Trial. JAMA Neurol. 2015 Jul;72(7):764-72. doi: 10.1001/jamaneurol.2015.0654. PMID 26010803
- [Result] Park KH, Jeong MH, Lee KH, Sim DS, Yoon HJ, Yoon NS, Kim KH, Park HW, Hong YJ, Kim JH, Ahn Y, Cho JG, Park JC, Kang JC. Comparison of peri-procedural platelet inhibition with prasugrel versus adjunctive cilostazol to dual anti-platelet therapy in patients with ST segment elevation myocardial infarction. J Cardiol. 2014 Feb;63(2):99-105. doi: 10.1016/j.jjcc.2013.07.004. Epub 2013 Sep 5. PMID 24012432
- [Result] Hwang G, Kim JG, Song KS, Lee YJ, Villavicencio JB, Suroto NS, Park NM, Park SJ, Jeong EA, Kwon OK. Delayed ischemic stroke after stent-assisted coil placement in cerebral aneurysm: characteristics and optimal duration of preventative dual antiplatelet therapy. Radiology. 2014 Oct;273(1):194-201. doi: 10.1148/radiol.14140070. Epub 2014 Jun 11. PMID 24918960
- [Derived] Ban SP, Kwon OK, Kim YD, Shim HS, Sung SB, Bang JS, Lee SU, Lee SH, Choi TW, Park Y. Comparison of Triple Antiplatelet (Aspirin, Clopidogrel, and Cilostazol) and Modified Dual Antiplatelet (Aspirin and Low-Dose Prasugrel) Therapy in Patients With High On-Treatment Platelet Reactivity Undergoing Stent-Assisted Coil Embolization for an Unruptured Intracranial Aneurysm: A Prospective Randomized Clinical Trial. Neurosurgery. 2025 Oct 10. doi: 10.1227/neu.0000000000003791. Online ahead of print. PMID 41070954